

IRAS number: 27844



## CONSENT FORM FOR PARTICIPANTS IN RESEARCH STUDIES - Online Screening

Please complete this form after you have read the Information Sheet.

<u>Title of Study:</u> SHAPER-PND: Community singing interventions for postnatal depression: a hybrid type II effectiveness-implementation trial

In order for us to then contact you if you are potentially eligible for our study, we would like to ask you to read this consent form.

Your information may be subject to review by responsible individuals from the research team for screening, monitoring and audit purposes.

Confidentiality will be maintained and you will not be identified in any research outputs.

| Please read the statements below and tick "yes" or "no". | Yes | No |
|---|---|---|
| 1. I consent to the processing of my personal information for the purposes of being contacted for the study. I understand that such information will be handled in accordance with the terms of the General Data Protection Regulation. | | |
| 2. I consent to my contact details being retained so that I may be invited to re-screen in the future, should I not be eligible to enrol in the study at this time based on my screening answers. | | |
| 3. I consent to my GP being contacted if there are any concerns for my or my baby's wellbeing. | | |

Thank you for reading the participant information sheet and the informed consent form. Please make sure you have ticket "yes" or "no" to be above points before submitting your personal information.



IRAS number: 278445



## **CONSENT FORM FOR PARTICIPANTS IN RESEARCH STUDIES**

Please complete this form after you have read the Information Sheet and/or listened to an explanation about the research.

<u>Title of Study:</u> SHAPER-PND: Community singing interventions for postnatal depression: a hybrid type II effectiveness-implementation trial

Thank you for considering taking part in this research. One of the researchers from the research team will explain the project to you before you agree to take part. If you have any questions arising from the Information Sheet or explanation already given to you, please ask the researcher before you decide whether you should join in. You will be given a copy of this Consent Form to keep and refer to at any time.

Your information may be subject to review by responsible individuals from the research team for screening, monitoring and audit purposes.

Confidentiality will be maintained and you will not be identified in any research outputs.

| | Yes | NO |
|---|---|---|
| I confirm that I understand that by ticking/initialling a 'Yes' box, I am consenting to being involved in this element of the study. I confirm that I understand that by ticking/initialling a 'No' box, I DO NOT consent to being involved in this element of the study. | | |
| 1. I confirm that I have read and understood the information sheet dated [INSERT DATE AND VERSION NUMBER] for the above study. I have had the opportunity to consider the information and asked questions which have been answered to my satisfaction. | | |
| 2. I consent voluntarily for myself and for my baby to be a participant in this study and understand that I can withdraw from the study at any time, without having to give a reason. | | |
| I consent to the processing of my personal information for the purposes explained to me in the Information Sheet. I understand that such information will be handled confidentially, in accordance with the terms of the General Data Protection Regulation. | | |
| I agree that the research team may use my data for future research within and outside the EU and understand that any such use of identifiable data would be reviewed and approved by a research ethics committee. In such cases, as with this project, data will not be identifiable in any report. | | |
| I agree to be contacted in the future by King's College London researchers who would like to invite me to participate in follow up studies to this project, or in future studies of a similar nature. | | |

Participant ICF Version 1.7 – 29-Sept-20

| | I agree to provide details of my GP and understand that if any safeguarding issues rise, my GP might be contacted to discuss the best way to support me and my baby. | |
|---|---|---|
| 7. I agree to record short videos being taken of play interaction in a comfortable setting between my baby and me. This recording aims to look at how me and my baby interact with each other and the information obtained can be used for our research. | | |
| 8. I agree to my views shared in focus groups and subsequent interviews to be recorded (in audio and/or video format) for data collection. The researchers may use a transcription service to transcribe the recordings into a different format. I understand that my identity will stay anonymous and I will not be identifiable in the published data or materials. (optional) | | |
| 9. I agree to provide biological samples (saliva and hair) throughout the study in accordance to the study protocol. These samples may be used for future studies and my data will remain anonymous. (optional) | | |
| 10. I agree to provide biological samples (saliva only) of my baby in accordance to the study protocol. These samples may be used for future studies and the data will remain anonymous. (optional) | | |
| 11. I agree to be contacted by implementation science researchers to provide my views on the study. I understand that my views may be video and audio recorded and published but I will not be identifiable in any of the research outputs. (optional) | | |
| 12. I do not wish to participate in the study, but I agree to be contacted by implementation science researchers for a brief interview, to explain why. (optional) | | |
| mandatory but are still ar | eent to points 1-7 in order<br>in integral part of the study.<br>ed to tell us why (optional), j | If you do not wish to pa |
| Participant: | | |
| Your Name | Date | Signature |
| Researcher: | | |
| Name of Researcher | Date | Signature |

IRAS number: 278445



IRAS number: 278445



## **CONSENT FORM FOR STAKEHOLDERS IN RESEARCH STUDIES**

Please complete this form after you have read the Information Sheet and/or listened to an explanation about the research.

<u>Title of Study:</u> SHAPER-PND: Community singing interventions for postnatal depression: a hybrid type II effectiveness-implementation trial

Thank you for considering taking part in this research. One of the researchers from the research team will explain the project to you before you agree to take part. If you have any questions arising from the Information Sheet or explanation already given to you, please ask the researcher before you decide whether you should join in. You will be given a copy of this Consent Form to keep and refer to

at any time.

| , | |
|---|---|
| Your information may be subject to review by responsible individuals from the research team for screening, monitoring and audit purposes. | |
| Confidentiality will be maintained and you will not be identified in any research outputs. | Yes No |
| I confirm that I understand that by ticking/initialling each 'Yes' box I am consenting to being involved in this element of the study. I understand that by ticking/initialling each 'No' box I DO NOT CONSENT to being involved in this element of the study. | |
| 1. I confirm that I have read and understood the information sheet dated [INSERT DATE AND VERSION NUMBER] for the above study. I have had the opportunity to consider the information and asked questions which have been answered to my satisfaction. | |
| 2. I consent voluntarily for myself to be a participant in this study and understand that I can withdraw from the study at any time, without having to give a reason. | |
| 3. I consent to the processing of my personal information for the purposes explained to me in the Information Sheet. I understand that such information will be handled in accordance with the terms of the General Data Protection Regulation. | |
| 4. I agree that the research team may use my data for future research within and outside the EU and understand that any such use of identifiable data would be reviewed and approved by a research ethics committee. In such cases, as with this project, data will not be identifiable in any report. | |
| 5. I agree that the research team may use my data for future research and understand that any such use of identifiable data would be reviewed and approved by a research ethics committee. In such cases, as with this project, data would not be identifiable in any report. | |
| 6. I agree to have my views recorded in focus groups and/or interviews. I am aware that my data will be anonymised, and I will not be identified in the published data. I understand that my views may be video and audio recorded and published but I will not be identifiable in any of the research outputs. | |

| Participant: | | |
|--------------|----------|-----------|
| Your Name | <br>Date | Signature |
| Researcher: | | |
| Name | Date | Signature |

Stakeholders ICF Version 1.5 – 30-Sep-20

IRAS number: 278445